CLINICAL TRIAL: NCT01468935
Title: Bone Marrow Cell Engraftment of the Uterus and Genetic Studies of Reproductive Functioning
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120016; 12-CH-0016
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-09-21

CONDITIONS: Endometriosis; Stem Cell Transplant; Healthy Volunteers
Keywords: Uterus; Endometrium; Bone Marrow Transplant; Gynecology; Healthy Volunteer; HV; Stem Cell Transplant; Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Some transplant recipients have been found to have cells in their uterus that come from the donor. Researchers want to study uterine tissue from three different groups of women: (1) healthy volunteers, (2) people who have had a stem cell transplant, and (3) people with rare diseases or conditions that affect reproduction. These samples will help researchers learn more about the way stem cells work in the reproductive tract.

Objectives:

- To collect cells from the uterus to study how stem cells work in the reproductive tract.

Eligibility:

- Women at least 18 years of age.

Design:

* Participants will be screened with a physical exam and medical history. They will also have blood and urine tests.
* Participants will have an endometrial biopsy to collect cells for study. The biopsy visit will take 1 to 2 hours.

DETAILED DESCRIPTION:
Transplantation with hematopoietic cells has been used for a wide variety of blood disorders, but also for diseases like solid organ cancers. Interestingly, women who have had bone marrow transplants have been found to have donor tissue in their endometrium, which raises the possibility of cellular therapies using bone marrow derived cells for gynecologic indications. Donor engraftment does not appear to occur when transplantations were performed with stem cells collected from peripheral blood of the donor. Therefore, the subtype of cells from the bone marrow responsible for engraftment is not yet known, nor is the ideal transplantation regimen known.

The immediate aim of this tissue procurement protocol is to obtain endometrial (uterine) stem cells from many human volunteers in order to examine the biological properties of those cells. We will collect tissue from 3 primary groups of patients: normal controls, patients with rare diseases or reproductive disorders, and patients who have undergone hematopoietic stem cell transplant. Each volunteer will undergo an endometrial biopsy during an office visit. The endometrial tissue will then be studied for a better understanding of their biological properties, growth and differentiation. One specific area of interest is to study how hematopoietic transplantation impacts endometrial cell function. These endometrial cells will be analyzed in-depth in the laboratory to determine if they came from the donor or recipient, and if so, which specific populations of cells. Hematologic pre-transplant conditioning information will be correlated with these research studies to identify factors that may assist with the understanding of adult endometrial stem cell biology.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subject is able to give consent/assent to participate in the protocol.

Listed below are acceptable medical conditions for inclusion in this protocol:

* Age greater than or equal to 18 years old
* Female gender
* Presence of a uterus
* Fall into one of the following categories:
* Healthy volunteers
* Hematologic patients:
* Whole bone marrow transplant recipients
* Peripheral blood stem cell transplant recipients
* Mesenchymal stem cell transplant recipients
* Bone marrow or stem cell donors
* Fully ablative transplant recipients
* Nonmyeloablative transplant recipients
* Cord blood transplant recipients

Rare, interesting, or unique reproductive phenotypes that may provide insight to endometrial function in health and disease:

* Asherman s syndrome
* Endometriosis
* Abnormal uterine bleeding
* Recurrent pregnancy loss
* Infertility
* Implantation failure
* Reproductive disorders

EXCLUSION CRITERIA:

* Unable to comprehend the investigational nature of the protocol participation.
* Positive pregnancy test.
* Anticoagulation or known coagulopathy.
* Active gonorrhea or Chlamydia infections or pelvic inflammatory disease within the last 3 months.
* Previous hysterectomy or endometrial ablation procedure.
* Thrombocytopenia (<50,000).
* Uterine or cervical cancer.
* Cervical stenosis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-10-31; Study Completion 2017-09-21

PRIMARY OUTCOMES:
To study if endometiral stem cells are different in normal and disease states.

SECONDARY OUTCOMES:
To study if the type of hematopoietic transplantation regimen affects uterine engraftment of donor stem cells.

CONTACTS AND LOCATIONS:
Overall Officials: Alan H DeCherney, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bhanu NV, Trice TA, Lee YT, Gantt NM, Oneal P, Schwartz JD, Noel P, Miller JL. A sustained and pancellular reversal of gamma-globin gene silencing in adult human erythroid precursor cells. Blood. 2005 Jan 1;105(1):387-93. doi: 10.1182/blood-2004-04-1599. Epub 2004 Sep 14. PMID 15367428
- [Background] Ogawa M, LaRue AC, Drake CJ. Hematopoietic origin of fibroblasts/myofibroblasts: Its pathophysiologic implications. Blood. 2006 Nov 1;108(9):2893-6. doi: 10.1182/blood-2006-04-016600. Epub 2006 Jul 13. PMID 16840726
- [Background] Taylor HS. Endometrial cells derived from donor stem cells in bone marrow transplant recipients. JAMA. 2004 Jul 7;292(1):81-5. doi: 10.1001/jama.292.1.81. PMID 15238594